CLINICAL TRIAL: NCT00943631
Title: A Phase II Study in Healthy Adult and Elderly Populations to Assess the Safety and Immunogenicity of an Unadjuvanted Sanofi Pasteur H1N1 Influenza Vaccine Administered at Two Dose Levels
Brief Title: Sanofi H1N1 Influenza Vaccine Administered at Two Dose Levels in Adult and Elderly Populations
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0053; N01AI80057C
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2011-04-13 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2010-03

CONDITIONS: Influenza
Keywords: H1N1, influenza A viruses, vaccine, elderly
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Group 2: H1N1 Vaccine 30 mcg (Experimental): 200 subjects (100 subjects ages 18-64 and 100 subjects greater than or equal to age 65) to receive 30 mcg of H1N1 vaccine on Days 0 and 21.
  Interventions: Biological: Inactivated H1N1 Vaccine
- Group 1: H1N1 Vaccine 15 mcg (Experimental): 200 subjects (100 subjects ages 18-64 and 100 subjects greater than or equal to age 65) to receive 15 mcg of H1N1 vaccine on Days 0 and 21.
  Interventions: Biological: Inactivated H1N1 Vaccine

INTERVENTIONS:
Biological: Inactivated H1N1 Vaccine — Two doses of inactivated influenza H1N1 vaccine delivered intramuscularly as 15 or 30 mcg per dose.

SUMMARY:
The purpose of this study is to assess the safety and the body's immune response (body's defense against disease) to an experimental H1N1 influenza vaccine in healthy adult and elderly populations. The study will enroll up to 450 healthy adults ages 18 and older with no history of H1N1 infection or vaccination. Two hundred individuals will be 18-64 years old, and the other 200 will be greater than or equal to 65 years of age. Participants will be randomly assigned to 1 of 2 possible vaccine groups: group 1 will receive 15 mcg of H1N1 vaccine; group 2 will receive 30 mcg of H1N1 vaccine. Both groups will receive vaccine injections on days 0 and 21 in the arm muscle. Study procedures include: medical history, physical exam, maintaining a memory aid, and blood sample collection. Participants will be involved in study related procedures for approximately 7 months.

DETAILED DESCRIPTION:
Recently, a novel swine-origin influenza A/H1N1 virus was identified as a significant cause of febrile respiratory illnesses in Mexico and the United States. It rapidly spread to many countries around the world, prompting the World Health Organization (WHO) to declare a pandemic on June 11, 2009. Data from several cohorts in different age groups that received licensed trivalent seasonal influenza vaccines suggest that these vaccines are unlikely to provide protection against the new virus. In addition, adults are more likely to have measurable levels of serum hemagglutination inhibition assay (HAI) or neutralizing antibody than are children. These data indicate the need to develop vaccines against the new H1N1 strain and suggest that different vaccine strategies (e.g., number of doses, need for adjuvant) may be appropriate for persons in different age groups. The primary safety objective of this study is to assess the safety of the unadjuvanted, inactivated H1N1 vaccine when administered at the 15 or 30 mcg dose. The primary immunogenicity objective is to assess the antibody response following a single dose of unadjuvanted, inactivated H1N1 vaccine, stratified by age of recipient, when administered at the 15 or 30 mcg dose. The secondary immunogenicity objective is to assess the antibody response following 2 doses of unadjuvanted, inactivated H1N1 vaccine, stratified by age of recipient, when administered at the 15 or 30 mcg dose. Participants will include up to 450 healthy adults age 18 and older who have no history of novel influenza H1N1 2009 infection or novel influenza H1N1 2009 vaccination. This is a randomized, double-blinded, Phase II study in healthy males and non-pregnant females designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 virus vaccine at 2 dose levels. Subjects will be randomized into 2 dose groups, stratified by age (200 subjects per dose group with 100 subjects per age stratum, 18-64 or greater than or equal to 65 years of age) to receive intramuscular influenza H1N1 vaccine at 15 mcg (Group 1) or 30 mcg (Group 2). The H1N1 vaccine will be administered at Day 0 and Day 21. Following immunization, safety will be measured by assessment of adverse events through 21 days following the last vaccination (Day 42 for those receiving both doses and Day 21 for those who do not receive the second dose), serious adverse events and new-onset chronic medical conditions through 7 months post first vaccination (Day 201), and reactogenicity to the vaccine for 8 days following each vaccination (Day 0-7). Immunogenicity testing will include HAI and neutralizing antibody testing on serum obtained on the day of each vaccination (prior to vaccination), on Day 8-10 after each vaccination, and 21 days following the second vaccination (Day 42).

ELIGIBILITY:
Inclusion Criteria:

* Are males or non-pregnant females age 18 and older, inclusive.
* Women of child-bearing potential (not surgically sterile via tubal ligation, bilateral oophorectomy or hysterectomy or who are not postmenopausal for greater than or equal to 1 year) must agree to practice adequate contraception that may include, but is not limited to, abstinence, monogamous relationship with vasectomized partner, barrier methods such as condoms, diaphragms, spermicides, intrauterine devices, and licensed hormonal methods during the study for at least 30 days following the last vaccination.
* Are in good health, as determined by vital signs, medical history to ensure any existing medical diagnoses or conditions are stable and not considered clinically significant, and targeted physical examination based on medical history. A stable chronic medical condition is defined as no change in prescription medication, dose, or frequency of medication in the last 3 months and health outcomes of the specific disease are considered to be within acceptable limits in the last 6 months. Any change that is due to change of health care provider, insurance company etc, or that is done for financial reasons, as long as in the same class of medication will not be considered a violation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome will not be considered a violation of this inclusion criterion.
* Are able to understand and comply with planned study procedures.
* Provide written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Have a known allergy to eggs or other components of the vaccine (including gelatin, formaldehyde, octoxinol, thimerosal, and chicken protein).
* Have a positive urine or serum pregnancy test within 24 hours prior to vaccination (if female of childbearing potential), or women who are breastfeeding.
* Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within the preceding 36 months.
* Have an active neoplastic disease or a history of any hematologic malignancy.
* Have long term use of glucocorticoids including oral, parenteral or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months. (Nasal and topical steroids are allowed.)
* Have a diagnosis of schizophrenia, bipolar disease, or other major psychiatric diagnosis.
* Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others, within the past 10 years.
* Are receiving psychiatric drugs (aripiprazole, clozapine, ziprasidone, haloperidol, molindone, loxapine, thioridazine, thiothixene, pimozide, fluphenazine, risperidone, mesoridazine, quetiapine, trifluoperazine, chlorprothixene, chlorpromazine, perphenazine, trifluopromazine, olanzapine, carbamazepine, divalproex sodium, lithium carbonate or lithium citrate). Subjects who are receiving a single antidepressant drug and are stable for at least 3 months prior to enrollment, without de-compensating symptoms will be allowed to be enrolled in the study.
* Have a history of receiving immunoglobulin or other blood product within the 3 months prior to vaccination in this study.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study or expect to receive an experimental agent during this study (prior to the Day 201 follow-up call - 180 days after the second vaccination).
* Have received any live licensed vaccines within 4 weeks or inactivated licensed vaccines within 2 weeks prior to vaccination in this study or plan receipt of such vaccines within 21 days following the second vaccination. This is inclusive of seasonal influenza vaccines.
* Have an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, or would interfere with the evaluation of responses.
* Have a history of severe reactions following previous immunization with influenza virus vaccines.
* Have an acute illness, including an oral temperature greater than 100.4 degrees Fahrenheit, within 3 days prior to vaccination.
* Have any condition that would, in the opinion of the site investigator, place them at an unacceptable risk of injury or render them unable to meet the requirements of the protocol.
* Participated in a novel influenza H1N1 2009 vaccine study in the past two years or have a history of novel influenza H1N1 2009 infection prior to enrollment.
* Have known active human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C infection.
* Have a history of alcohol or drug abuse in the last 5 years.
* Plan to travel outside of North America in the time between the first vaccination and 42 days following the first vaccination.
* Have a history of Guillain-Barré Syndrome.
* Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Duke Translational Medicine Institute - Clinical Vaccine Unit, Durham, North Carolina
  - Vanderbilt University - Pediatric - Vanderbilt Vaccine Research Center, Nashville, Tennessee

REFERENCES:
- [Result] Chen WH, Winokur PL, Edwards KM, Jackson LA, Wald A, Walter EB, Noah DL, Wolff M, Kotloff KL; Pandemic H1N1 Vaccine Adult Study Group. Phase 2 assessment of the safety and immunogenicity of two inactivated pandemic monovalent H1N1 vaccines in adults as a component of the U.S. pandemic preparedness plan in 2009. Vaccine. 2012 Jun 13;30(28):4240-8. doi: 10.1016/j.vaccine.2012.04.044. Epub 2012 Apr 23. PMID 22537984

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adult males and females recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled and vaccinated between 07AUG2009 and 18AUG2009.
Groups:
- H1N1 Vaccine 15 Mcg: Participants received 15 mcg of H1N1 vaccine by intramuscular injection on Days 0 and 21.
- H1N1 Vaccine 30 Mcg: Participants received 30 mcg of H1N1 vaccine by intramuscular injection on Days 0 and 21.
Period: Overall Study
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Started | 202 | 204
Completed | 198 | 202
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg | Total
Number analyzed (Participants) | 202 | 204 | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 100 | 202
  >=65 years | 100 | 104 | 204
Age Continuous [Mean (Standard Deviation); unit: years] | 58.7 (17.1) | 59.6 (16.4) | 59.1 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 112 | 215
  Male | 99 | 92 | 191
Region of Enrollment [Number; unit: participants]
  United States | 202 | 204 | 406

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Vaccine-associated Serious Adverse Events (SAEs)
Description: Serious adverse events included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required in-patient hospitalization or prolongation thereof; resulted in a congenital anomaly/birth defect; or may have jeopardized the participant or required intervention to prevent one of these outcomes. Association to vaccination was determined by a study clinician licensed to make medical diagnoses.
Time Frame: Day 0 through Day 180 after last vaccination
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 202 | 204
Participants | 0 | 0

2. Primary Outcome: Number of Participants Reporting Solicited Local Reactions Based on the Functional Grading Scale After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of pain, tenderness and swelling for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 202 | 204
Participants
  Pain | 36 | 34
  Tenderness | 58 | 75
  Swelling | 27 | 16

3. Primary Outcome: Number of Participants Reporting Solicited Local Reactions Based on the Functional Grading Scale After the Second Vaccination
Description: as for outcome 2
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 192 | 197
Participants
  Pain | 27 | 27
  Tenderness | 54 | 63
  Swelling | 10 | 18

4. Primary Outcome: Number of Participants Reporting Measured Injection Site Reactions of Swelling and Redness After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of local reactions of swelling and redness for 8 days after vaccination (Day 0-7). If the reaction was present, the maximum diameter was measured in millimeters (mm). Participants are counted if they reported experiencing the reaction with any measurement greater than 0 mm on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 202 | 204
Participants
  Swelling | 31 | 22
  Redness | 39 | 32

5. Secondary Outcome: Number of Participants in the 18-64 Year Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 8-10 and 21 Days Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants prior to the initial vaccination as well as 8-10 and 21 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post vaccination 2 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 post vaccination 2 titer was an increase by 4-fold or more.
Time Frame: Baseline and Day 8-10 and 21 after the second vaccination
Population: Participants were included in the analyses if they received the both vaccinations and had blood collected at the timepoints. Participants were analyzed as treated. This outcome measure restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 95 | 95
Participants
  Day 8-10 | 86 | 83
  Day 21 | 84 | 82

6. Secondary Outcome: Number of Participants in the 65 Years and Older Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 8-10 Days Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants prior to the initial vaccination and 8-10 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post vaccination 2 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 post vaccination 2 titer was an increase by 4-fold or more.
Time Frame: Baseline and Day 8-10 after the second vaccination
Population: Participants were included in the analyses if they received the both vaccinations and had blood collected at the timepoints. Participants were analyzed as treated. This outcome measure restricts to age stratum. One subject was excluded due to receipt of a non-study vaccine prior to the clinic visit.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 94 | 100
Participants | 68 | 84

7. Primary Outcome: Number of Participants Reporting Measured Injection Site Reactions of Swelling and Redness After the Second Vaccination
Description: as for outcome 4
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 192 | 197
Participants
  Swelling | 11 | 18
  Redness | 33 | 25

8. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactions Based on the Functional Grading Scale After the First Vaccination
Description: Participants maintained a memory aid to record daily the occurrence of systemic symptoms of feverishness, malaise, myalgia, headache, and nausea for 8 days after vaccination (Day 0-7) based on their interference with daily activities. Participants are counted if they reported experiencing the symptom at any severity on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 202 | 204
Participants
  Feverishness | 11 | 5
  Malaise | 31 | 30
  Myalgia | 23 | 22
  Headache | 46 | 42
  Nausea | 5 | 6

9. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactions Based on the Functional Grading Scale After the Second Vaccination
Description: as for outcome 8
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 192 | 197
Participants
  Feverishness | 11 | 10
  Malaise | 32 | 25
  Myalgia | 25 | 18
  Headache | 20 | 33
  Nausea | 10 | 11

10. Primary Outcome: Number of Participants Reporting Fever After the First Vaccination
Description: Participants were provided with a thermometer and a memory aid on which to record daily oral temperatures for 8 days after vaccination (Day 0-7). The protocol defined fever as oral temperature of 38.0 degrees Celsius or higher. Participants are counted as experiencing fever if they reported oral temperatures of 38.0 degrees Celsius or higher on any of the 8 days.
Time Frame: Day 0-7 after first vaccination
Population: All participants receiving the first vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 202 | 204
Participants | 2 | 1

11. Primary Outcome: Number of Participants Reporting Fever After the Second Vaccination
Description: as for outcome 10
Time Frame: Day 0-7 after second vaccination
Population: All participants receiving the second vaccination are included in the safety ITT cohort.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 192 | 197
Participants | 2 | 0

12. Primary Outcome: Number of Participants in the 18-64 Year Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 8-10 Days Following 1 Dose of Vaccine
Description: Blood was collected from all participants prior to vaccination and at the 8-10 day follow up visit for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 8-10 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 8-10 titer was an increase by 4-fold or more.
Time Frame: Baseline and Day 8-10 after first vaccination
Population: Participants were included in the analyses if they received the first vaccination and had blood collected at both timepoints. Participants were analyzed as treated. This outcome measure restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 101 | 100
Participants | 80 | 85

13. Primary Outcome: Number of Participants in the 65 Years and Older Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 8-10 Days Following 1 Dose of Vaccine
Description: as for outcome 12
Time Frame: Baseline and Day 8-10 after first vaccination
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 100 | 104
Participants | 63 | 69

14. Primary Outcome: Number of Participants in the 18-64 Year Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 21 Days Following 1 Dose of Vaccine
Description: Blood was collected from all participants prior to vaccination and at the 21 day follow up visit for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 8-10 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 8-10 titer was an increase by 4-fold or more.
Time Frame: Baseline and Day 21 after first vaccination
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 100 | 98
Participants | 86 | 87

15. Primary Outcome: Number of Participants in the 65 Years and Older Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 21 Days Following 1 Dose of Vaccine
Description: as for outcome 14
Time Frame: Baseline and Day 21 after first vaccination
Population: Participants were included in the analyses if they received the first vaccination and had blood collected at both timepoints. Participants were analyzed as treated. This outcome measure restricts to age stratum. One participant was excluded due to the blood being collected after administration of the second vaccination.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 98 | 103
Participants | 66 | 83

16. Primary Outcome: Number of Participants in the 18-64 Year Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus Prior to and at 8-10 Days Following 1 Dose of H1N1 Vaccine
Description: Blood was collected from all participants prior to vaccination and at the 8-10 day follow up visit for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 0 prior to and Day 8-10 after first vaccination
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 101 | 100
Participants
  Day 0 | 14 | 9
  Day 8 | 85 | 89

17. Secondary Outcome: Number of Participants in the 65 Years and Older Age Stratum With 4-fold or Greater HAI Antibody Titer Increases Against Influenza H1N1 2009 Virus at 21 Days Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants prior to the initial vaccination and 21 days after the second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. A participant met the threshold of a 4-fold rise in titer if the Day 0 titer was less than 1:10 (the assay's lowest level of detection) and the Day 21 post vaccination 2 titer was 1:40 or greater, or the Day 0 titer was greater than or equal to 1:10 and the Day 21 post vaccination 2 titer was an increase by 4-fold or more.
Time Frame: Baseline and Day 21 after the second vaccination
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 95 | 101
Participants | 70 | 82

18. Secondary Outcome: Number of Participants in the 18-64 Year Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus at 8-10 and 21 Days Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants at Day 8-10 and Day 21 post second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 8-10 and Day 21 after the second vaccination
Population: Participants were included in the analyses if they received both vaccinations and had blood collected at the timepoints. Participants were analyzed as treated. This outcome measure restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 95 | 95
Participants
  Day 8-10 | 88 | 86
  Day 21 | 88 | 87

19. Primary Outcome: Number of Participants in the 65 Years and Older Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus Prior to and at 8-10 Days Following 1 Dose of H1N1 Vaccine
Description: as for outcome 16
Time Frame: Day 0 prior to and Day 8-10 after first vaccination
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 100 | 104
Participants
  Day 0 | 24 | 25
  Day 8 | 80 | 84

20. Primary Outcome: Number of Participants in the 18-64 Year Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus at 21 Days Following 1 Dose of H1N1 Vaccine
Description: Blood was collected from all participants at the 21 day follow up visit for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after first vaccination
Population: Participants were included in the analyses if they received the first vaccination and had blood collected at the timepoint. Participants were analyzed as treated. This outcome measure restricts to age stratum.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 100 | 98
Participants | 90 | 90

21. Primary Outcome: Number of Participants in the 65 Years and Older Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus at 21 Days Following 1 Dose of H1N1 Vaccine
Description: as for outcome 20
Time Frame: Day 21 after first vaccination
Population: Participants were included in the analyses if they received the first vaccination and had blood collected at the timepoint. Participants were analyzed as treated. This outcome measure restricts to age stratum. One participant was excluded due to the blood being collected after administration of the second vaccination.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 98 | 103
Participants | 79 | 94

22. Secondary Outcome: Number of Participants in the 65 Years and Older Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus at 8-10 Days Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants at Day 8-10 post second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 8-10 after the second vaccination
Population: Participants were included in the analyses if they received both vaccinations and had blood collected at the timepoint. Participants were analyzed as treated. This outcome measure restricts to age stratum. One subject was excluded due to receipt of an non-study vaccine prior to the clinic visit.
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 94 | 100
Participants | 80 | 92

23. Secondary Outcome: Number of Participants in the 65 Years and Older Age Stratum With a Serum Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater Against Influenza H1N1 2009 Virus at 21 Days Following 2 Doses of H1N1 Vaccine
Description: Blood was collected from all participants at Day 21 post second vaccination for testing in the HAI assay with Influenza H1N1 2009 virus as the assay antigen. Each sample was tested at least twice according to standard operating procedures and the result of each replicate reported. A participant is counted if the geometric mean of the replicate values was 1:40 or greater.
Time Frame: Day 21 after the second vaccination
Population: as for outcome 22
Measure: Number; unit: Participants
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Number analyzed (Participants) | 95 | 101
Participants | 79 | 93

ADVERSE EVENTS:
Time Frame: Solicited events were collected for 8 days after each vaccination, unsolicited events through 21 days after last vaccination, and serious adverse events and new onset chronic medical conditions through 180 days after last vaccination.
Description: For events solicited on a Memory Aid in the 8 days after vaccination, a participant was considered to have one event if it was reported as experienced at any time in the 8 day period.
Arm/Group | H1N1 Vaccine 15 Mcg | H1N1 Vaccine 30 Mcg
Serious Adverse Events (participants affected / at risk) | 6/202 | 5/204
Other Adverse Events (participants affected / at risk) | 149/202 | 150/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H1N1 Vaccine 15 Mcg (N=202) | H1N1 Vaccine 30 Mcg (N=204)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Thoracotomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H1N1 Vaccine 15 Mcg (N=202) | H1N1 Vaccine 30 Mcg (N=204)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 10 (10)
Feeling hot (General disorders) | 21 (22) | 14 (15)
Malaise (General disorders) | 54 (63) | 48 (55)
Myalgia (Musculoskeletal and connective tissue disorders) | 42 (48) | 34 (40)
Headache (Nervous system disorders) | 57 (66) | 59 (75)
Nausea (Gastrointestinal disorders) | 13 (15) | 17 (17)
Injection site pain (General disorders) | 49 (63) | 48 (61)
Tenderness (General disorders) | 86 (112) | 94 (138) — Tenderness was solicited as a reaction at the vaccination site.
Injection site erythema (General disorders) | 57 (72) | 42 (57)
Injection site swelling (functional grading) (General disorders) | 31 (37) | 29 (34) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.
Injection site swelling (measured) (General disorders) | 36 (42) | 35 (40) — Injection site swelling was solicited separately for functional grading of impact on daily activities and as a measured reaction.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less